CLINICAL TRIAL: NCT00421577
Title: Usage of Laboratory Technique for Localization of Caries Associated Bacteria on Tooth Surfaces as Clinical Measurement to Caries Diagnosis and Treatment Efficiency.
Brief Title: Technique for Localization of Caries Associated Bacteria on Tooth Surfaces.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: gum-HMO-CTIL
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2007-01-12 (Estimated); Status verified 2007-01

CONDITIONS: Caries
Keywords: Caries Diagnosis; Replica technique

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
There is a simple laboratory technique for localization of caries associated bacteria on tooth surfaces by taking an impression of the teeth with a material containing sucrose.

The purpose of this study is to check whether the technique can be incorporated into dental clinics as diagnostic tool comparing to other diagnostic methods available.

ELIGIBILITY:
Inclusion Criteria:

* adult/ patient of the student clinic in Hadassa, Jerusalem.

Exclusion Criteria:

* children/ antibiotic taken in the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shay Levi, DMD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Result] Rosenberg M, Weiss E, Eli I. A novel replica technique for localization of caries-associated bacteria on tooth surfaces: development and initial experience. Caries Res. 1988;22(1):42-4. doi: 10.1159/000261081. No abstract available. PMID 3275501